CLINICAL TRIAL: NCT04830501
Title: A Phase I Study of the Safety, Tolerability, Pharmacokinetics Profile, and Preliminary Efficacy of TT-00434 in Patients With Advanced Solid Tumors
Brief Title: Study of the of the Safety and Tolerability of TT-00434 in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: TransThera Sciences (Nanjing), Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TT00434CN01
Record Dates: First submitted 2021-03-28; First posted 2021-04-05 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose Escalation (Experimental): This study adopts an accelerated titration design (ATD) and utilizes an accelerated dose escalation phase in order to minimize suboptimal drug exposures, followed by a conventional 3+3 dose escalation phase to achieve MTD.
  Interventions: Drug: TT-00434

INTERVENTIONS:
Drug: TT-00434 — Once daily [QD], 28 days/cycle.

SUMMARY:
This is a phase I study of the safety, tolerability, pharmacokinetics profile, and preliminary efficacy of TT-00434 in patients with advanced solid tumors.

DETAILED DESCRIPTION:
This is a phase I, First-in-Human (FIH), open-label, dose escalation clinical study in patients who have a histological or cytologically confirmed diagnosis of advanced or recurrent tumors that all standard treatments have been used or are not feasible. It aims to determine the maximum tolerated dose (MTD) and/or the recommended phase 2 dose (RP2D) for study, evaluate the safety, tolerability, pharmacokinetic (PK) and pharmacodynamic (PD) characteristics and the preliminary anti-tumor activity of TT-00434, and explore the relationship between the anti-tumor activity of TT-00434 and the tumor FGFR alterations.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 20 years.
* Patients must have a histological or cytologically confirmed diagnosis of advanced or recurrent malignant solid tumors.
* Patients have received all currently available standard treatments (unless the therapy is contraindicated, intolerable or unavailable due to any reasons).
* Patients must have measurable or evaluable disease (according to RECIST 1.1)
* Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 2
* Must agree to take sufficient contraceptive methods to avoid pregnancy during the study and until at least 6 months after ceasing study treatment
* Patients must have fully understood and voluntarily signed informed consent form (ICF) for this study.

Exclusion Criteria:

* Patients who received other investigational products or devices in other clinical trials within 4 weeks before the first dose.
* Patients who received anti-tumor therapy within 4 weeks, or within 5-half-lives (which is longer) before the first dose, including but not limited to chemotherapy, radiotherapy (palliative radiotherapy is completed at least 2 weeks before the first dose can enrol), targeted therapy or immunotherapy.
* Patients who have previous toxicity of anti-tumor therapy that has not recovered to Grade 1. (except for ≤ Grade 2 alopecia, chemotherapy-induced peripheral neurotoxicity, and ototoxicity).
* Patients who have gastrointestinal disorders that will affect oral administration or the Investigator judges that the absorption of TT-00434 will be interfered.
* Patients underwent major surgery (except biopsy) within 4 weeks, or the surgical incision has not completely healed prior to the first dose.
* Patients who have active bacterial or fungal infections (CTCAE, Grade ≥ 2) that required systemic treatment within 2 weeks prior to the first dose.
* Patients who have active HBV infection (HBV DNA copies ≥ ULN) and/or HCV infection (HCV RNA copies ≥ ULN)
* Patients who test positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome.
* Has received a live-virus vaccination within 30 days of planned first dose NOTE: Seasonal flu vaccines are permitted.
* Known or suspected drug hypersensitivity to any ingredients of TT-00434 tablets.
* Female patients in pregnancy or lactation. Male patients or female patients at reproductive ages who are unwilling to receive effective contraceptive measures.
* Patients who are judged by the Investigator to be unsuitable for this study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2021-07-12 (Actual); Primary Completion 2023-10-18 (Actual); Study Completion 2023-10-18 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (DLT) | At the end of Cycle 1 (each cycle is 28 days)
  Safety and tolerability
Incidence of AEs | up to 30 days from study discontinuation
  Safety and tolerability

SECONDARY OUTCOMES:
Peak Plasma Concentration (Cmax) | At the end of Cycle 1 (each cycle is 28 days)
  PK evaluation
Area under the plasma concentration versus time curve (AUC) | At the end of Cycle 1 (each cycle is 28 days)
  PK evaluation
Time of first Occurance of Cmax（tmax) | At the end of Cycle 1 (each cycle is 28 days)
  PK evaluation
Serum phosphate levels | up to 30 days from study discontinuation
  PD biomarker
Objective response rate (ORR) | through study completion, an average of 1 year
  Assess anti-tumor activity
Disease control rate (DCR) | through study completion, an average of 1 year
  Assess anti-tumor activity
Progression Free Survival (PFS) | through study completion, an average of 1 year
  Assess anti-tumor activity
Overall Survival (OS) | through study completion, an average of 1 year
  Assess anti-tumor activity

CONTACTS AND LOCATIONS:
Overall Officials: Huey En Tzeng, Principal Investigator — Taipei Medical University Hospital; Chia Jui Yen, Principal Investigator — National Cheng-Kung University Hospital; Ching Liang Ho, Principal Investigator — Tri-Service General Hospital; Ming Che Liu, Principal Investigator — Taipei Medical University Hospital
Locations (3):
- Taiwan (3):
  - National Cheng Kung University Hospital, Tainan
  - Taipei Medical University Hospital, Taipei
  - Tri-Service General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No